CLINICAL TRIAL: NCT06556030
Title: Botulinum Toxin in Open Abdomen Closure
Brief Title: A Multicentre, Randomised, Single-blind, Controlled Protocol to Evaluate the Efficacy of Early Administration of Botulinum Toxin for Primary Midline Closure in Patients With Open Abdomen.
Acronym: BOTU-CLOSURE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOTU-CLOSURE
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-05

CONDITIONS: Botulinum Toxin Type A; Open Abdomen; Abdominal Wall; Clinical Trial
Keywords: botulinum toxin, open abdomen, laparostomy, abdominal wall closure, clinical trial.
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): physiological saline 50 cc
  Interventions: Other: CONTROL
- botulinum toxin (Experimental): Intramuscular injection into the flat muscles of the abdominal wall of 300/500 Units of botulinum toxin A dissolved in 100 cc of physiological saline, distributed in 5 points on each side of the abdomen in the first 48 hours after leaving the abdomen open.
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Botulinum Toxin
  Arms: botulinum toxin
Other: CONTROL — Saline Solution
  Arms: Control

SUMMARY:
A multicentre, randomised, single-blind, controlled protocol to evaluate the efficacy of early administration of botulinum toxin for primary midline closure in patients with open abdomen. Early use (less than 48 hours) of botulinum toxin as a neuromuscular abdominal wall blocker in patients whose abdomen is left open, regardless of the cause, will improve postoperative outcome and prognosis, leading to significantly higher percentages of primary midline closure.

DETAILED DESCRIPTION:
According to the definition of the World Society for Emergency Surgery (WSES), an open abdomen is defined as the intentional creation of a laparostomy by non-approximation of the aponeurotic edges of the rectus abdominis muscles in the midline (1). This technique is restricted to very specific situations, usually in the critically ill patient who has undergone damage control surgery for polytrauma, abdominal sepsis or abdominal compartment syndrome. In this context, it may be necessary to keep the abdomen open for four indications that were defined in 2015 by an international consensus of experts:

need for reintervention (second-look) in cases of ischaemia or severe intra-abdominal contamination; inability to close due to visceral oedema; traumatic damage to the abdominal wall; failure of medical treatment in the management of abdominal compartment syndrome (2).

Since its description in 1993 (although open abdomen was used for abdominal compartment syndrome decades earlier), the use of damage control surgery associated with intensive resuscitation has decreased mortality in these patients from 90% to approximately 20-30% today (3).

Despite its benefits for the survival of unstable patients, the creation of an open abdomen creates a non-anatomical situation with significant physiological repercussions: exposure of the abdominal viscera to the environment without barrier mechanisms results in hypothermia, and significant fluid and protein loss, precipitating a catabolic state that feeds back into the multi-organ failure of the critically ill patient. In addition, the open abdomen leads to potentially very serious complications such as the development of an enteroatmospheric fistula, which occurs in up to 15% of these patients (2,4,5).

In order to reduce complications and simplify the management of patients with open abdomen, various temporary closure devices have been developed (5). Among them, current evidence recommends the use of negative pressure devices, generally consisting of: a sheet of non-absorbable plastic material in contact with the viscera that tries to prevent the appearance of adhesions and fistulas and which, by presenting small perforations, allows intra-abdominal fluid to escape, a macroporous material that remains in lateral contact with the fascia and subcutaneous tissue, and a final occlusive cover to which suction is applied to generate the negative pressure. The incorporation of these devices has been shown to reduce the production of proinflammatory cytokines in the peritoneal fluid (6) and the aforementioned guidelines recommend their use in all cases of open abdomen (grade of recommendation B, level of evidence I)(2).

However, no temporary closure technique to date has been able to restore the physiological situation altered by having an open abdomen, and therefore all efforts should be directed towards keeping the duration of the open abdomen as short as possible.

There is a direct relationship between the duration of the open abdomen and the number of dressings or revisions required until closure, and the appearance of complications such as enteroatmospheric fistula (7). Although some temporary closure techniques can lengthen this time until the appearance of fistulas, it is generally established that the risk of fistula is very high after one week of open abdomen (8).

Another negative effect of open abdomen occurs at the level of the abdominal wall: as there is no continuity of the wall, the lateral musculature of the abdominal wall (external, internal and transverse oblique muscles) is functionally "disinserted" from its insertion in the midline, and naturally tends to retract as time goes by, thus separating the rectus abdominis muscles and hindering the eventual reconstruction of the midline when the patient's situation allows it.

In order to achieve greater primary fascial closure, various techniques have been described in association with temporary closures to prevent muscle retraction. The most common form is the interposition between the temporary closure materials of sutures or meshes anchored to both fascial ends. This not only prevents retraction, but in successive revision surgeries the tension on the musculature can be progressively increased to achieve closure after a few days. This is known as sequential closure or delayed primary closure, as the duration until complete closure is achieved is usually longer than 7 days, generally around 13-15 (4,9).

Another resource available to achieve fascial closure is to associate component separation techniques, commonly anterior component separation. However, these manoeuvres are associated with greater complications at the abdominal wall level such as haematoma formation. The third way would be to suture both ends of the fascia to a mesh that would be interposed between them containing the viscera, which in the literature has been called bridging, generally with a resorbable mesh. The subsequent occurrence of an eventration is greater than 50%, but it allows the abdominal wall to be closed and the defect to be addressed in a planned manner at a later date (10).

In summary, making the decision to leave an open abdomen is a race against time in which the longer it takes for the patient's clinical situation to allow closure, the more complications can occur, and the more difficult it is to achieve repair. The literature describes highly variable rates of primary fascial closure, with the best results being the combination of vacuum devices associated with traction techniques, with rates of up to 80% (11,12). Even within the same multicentre study with a closure rate of 65.5%, the range among participating centres was 25.5% to 85.2% (13). It should also be noted that these patients have a high risk of subsequent eventration with published rates of 35% at 4 years (14). Closure at the first surgical revision is achieved in only one third of patients, but these patients have fewer complications (15).

Botulinum toxin is a bacterial neurotoxin (Cl. botulinum) responsible for botulism. There are eight varieties of neurotoxin, all of which share the same mechanism of action: blocking the release of acetylcholine at the motor plate at the neuromuscular junction, generating a chemical denervation that is reversible. Medical applications have been described since the last decades of the last century.

of botulinum toxin infiltration for the treatment of muscle dystonia and also for aesthetic purposes (16).

In abdominal wall surgery, the use of botulinum toxin was first described in 2009 (17). As mentioned, its effect is reversible, becoming noticeable in experimental studies after 1-2 days, reaching a maximum after 3-4 weeks, and disappearing after 6-9 months. Due to this dynamic, its application has been mainly in the context of elective surgery in patients with large hernia defects, infiltrating the lateral musculature weeks before the operation. In this field, there are publications with good quality evidence (18) that support its use in patients with large eventrations and loss of domicile, alone or in combination with progressive pneumoperitoneum (19).

In the context of open abdomen and damage control surgery, the time to onset of significant paralysis and the clinical situation of the patients, which guides the timing and indication for reinterventions, have been the main factors limiting its applicability. The first mention of this indication was found in 2013 by Zielinski's group, who published a series of 18 patients who underwent infiltration with 300 IU of BTX in the external, internal and transverse oblique of the abdomen bilaterally. Primary fascial closure was achieved in 83%, bridging in another 6% and skin closure and formation of a planned eventration in 11%. Subsequent complications included 11% early dehiscence (20). However, in 2016, the same group published a pilot clinical trial in which the use of botulinum toxin did not significantly differ from the placebo group. This clinical trial had very restrictive exclusion criteria and consequently obtained primary closure figures with and without the use of toxin of over 90% that do not correspond to those described in other studies, which in the words of the authors themselves suggests a possible type II error (21). In addition to these studies, there are retrospective case series that provide favourable data without showing an increase in complications (22). All this is summarised in the systematic review of the literature published in 2022 (23): the use of botulinum toxin seems to offer advantages in the context of the open abdomen, without a high risk profile, although quality studies are needed to provide information on effectiveness based on a population that is more representative of reality.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must be able to understand the purpose and risks of the study, giving informed consent and authorising the use of confidential health information. If the patient is unable to consent due to emergency status, a first or second degree relative will be requested. If the patient recovers, the patient's consent to continue participation will be sought again.

  2. Subjects Patients over 18 years of age who, regardless of the cause, have undergone abdominal surgery, after which it has been necessary to leave the abdomen open.

  3. Subjects able and willing to participate and to be followed for most of the duration of the study.

Exclusion Criteria:

* Personal historyDiseases which, in the opinion of the investigator, may interfere with or worsen the action of the botulinum toxin. For example, patients with: hyperthyroidism, neuromuscular disease, myasthenia gravis, Eaton Lamber syndrome or ALS are excluded.

  2. Drugs that affect muscle tone or the autonomic nervous system, e.g. administration of antibiotics such as aminoglycosides, lincosamides, polymyxins or tetracyclines.

  3. Pregnancy or lactation. 4. Known hypersensitivity. 5. Active neoplastic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Main Endpoint | 30 days
  Percentage of patients achieving primary midline closure in the experimental group compared to the control group (within 20 days after the first procedure where the abdomen is left open).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Vaello Jodra, Consultant, Principal Investigator — Hospital Universitario del Henares; Luis Asensio Gomez, Consultant, Principal Investigator — Hospital Universitario La Paz

IPD SHARING:
Plan to Share IPD: Undecided